CLINICAL TRIAL: NCT01759212
Title: Safety and Efficacy of Intramyocardial Implantation of Allogeneic Mesenchymal Stem Cells in Patients With End-stage Heart Failure Undergoing Left Ventricular Assist Device Implantation
Brief Title: Left Ventricular Assist Device Combined With Allogeneic Mesenchymal Stem Cells Implantation in Patients With End-stage Heart Failure.
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of eligible patients
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Kyriakos Anastasiadis, Professor Kyriakos Anastasiadis, AHEPA University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEPA_CTL_02
Record Dates: First submitted 2012-12-18; First posted 2013-01-03 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure; Ischemic Cardiomyopathy
Keywords: stem cell implantation; coronary artery disease; left ventricular assist device
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem cells implantation (Experimental): Patients with end-stage heart failure due to ischemic cardiomyopathy will undergo combined cellular and mechanical support with implantation of off-the-shelf allogeneic mesenchymal stem cells and left ventricular assist device.
  Interventions: Biological: Allogeneic stem cells implantation

INTERVENTIONS:
Biological: Allogeneic stem cells implantation

SUMMARY:
The aim of the study is to investigate safety and efficacy of intramyocardial implantation of allogeneic mesenchymal stem cells in patients with end-stage ischemic cardiomyopathy undergoing left ventricular assist device implantation.

DETAILED DESCRIPTION:
End-stage ischemic cardiomyopathy (ICM) with non-graftable coronary arteries is a common and debilitating problem. The ultimate therapeutic goal in such cases is cardiac transplantation which is restricted by donor availability. Alternatively, left ventricular assist devices (LVAD) are increasingly used as bridge to transplantation or more recently as destination therapy in non-transplant candidates. Widely used second- and third-generation continuous-flow LVAD offer symptomatic relief and prolong life. However, LV unloading rarely improves native heart function in ischemic hearts. We aim to increase myocardial viability and improve native cardiac function in patients with end-stage ICM by injecting allogeneic bone marrow stem cells at the time of LVAD implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* End-stage heart failure due to ischemic cardiomyopathy that requires mechanical support according to current indications
* Ability to provide informed consent

Exclusion Criteria:

* Not willing to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Improvement in myocardial perfusion/viability | 12 months
  Improvement in myocardial perfusion/viability assessed with SPECT segmental analysis
Improvement in myocardial perfusion/viability | 24 months
  Improvement in myocardial perfusion/viability assessed with SPECT segmental analysis

SECONDARY OUTCOMES:
Morbidity | 12 months
  Major adverse cardiac and cerebrovascular events
Change in left ventricular function | one year
  Change in left ventricular function after combined mechanical and cellular therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, MD, PhD, FETCS, Principal Investigator — AHEPA University Hospital
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Anastasiadis K, Antonitsis P, Doumas A, Koliakos G, Argiriadou H, Vaitsopoulou C, Tossios P, Papakonstantinou C, Westaby S. Stem cells transplantation combined with long-term mechanical circulatory support enhances myocardial viability in end-stage ischemic cardiomyopathy. Int J Cardiol. 2012 Mar 22;155(3):e51-3. doi: 10.1016/j.ijcard.2011.07.062. Epub 2011 Aug 17. No abstract available. PMID 21852003
- [Background] Anastasiadis K, Antonitsis P, Argiriadou H, Koliakos G, Doumas A, Khayat A, Papakonstantinou C, Westaby S. Hybrid approach of ventricular assist device and autologous bone marrow stem cells implantation in end-stage ischemic heart failure enhances myocardial reperfusion. J Transl Med. 2011 Jan 19;9:12. doi: 10.1186/1479-5876-9-12. PMID 21247486
- [Background] Ibrahim M, Rao C, Athanasiou T, Yacoub MH, Terracciano CM. Mechanical unloading and cell therapy have a synergistic role in the recovery and regeneration of the failing heart. Eur J Cardiothorac Surg. 2012 Aug;42(2):312-8. doi: 10.1093/ejcts/ezs067. Epub 2012 Feb 29. PMID 22378852